CLINICAL TRIAL: NCT03643627
Title: A Phase 1a, Double-Blind, Placebo-Controlled, Single-Ascending Dose Study of SYNT001 in Healthy Volunteers
Brief Title: A Study of SYNT001 in Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Syntimmune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYNT-101
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Healthy
MeSH Terms: interventions — orilanolimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 1 mg/kg (Experimental)
  Interventions: Drug: SYNT001
- 3 mg/kg (Experimental)
  Interventions: Drug: SYNT001
- 10 mg/kg (Experimental)
  Interventions: Drug: SYNT001
- 30 mg/kg (Experimental)
  Interventions: Drug: SYNT001

INTERVENTIONS:
Drug: SYNT001 — single IV infusion
  Arms: 1 mg/kg; 10 mg/kg; 3 mg/kg; 30 mg/kg
Drug: Placebo — single IV infusion
  Arms: Placebo

SUMMARY:
This study is being done to compare the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of an intravenous (IV) formulation of SYNT001. This is the first-in-human (FIH) study of SYNT001.

ELIGIBILITY:
IInclusion Criteria:

Subjects must meet the following criteria to be included:

* Healthy as determined by comprehensive clinical assessment and clinical laboratory investigations
* Body mass index 18.5 to 30.0 kg/m2
* Must use medically acceptable contraception
* Willingness to complete all study measurements and assessments in compliance with the protocol

Exclusion Criteria:

Subjects meeting any of the following criteria are to be excluded:

* Past or present disease that is judged by the investigator to have the potential to interfere with the study procedures, compromise safety or affect the PK evaluations
* Subject unable or unwilling to comply with the protocol
* Any exposure to an investigational drug within the 30 days prior to screening
* Use of any tobacco or nicotine-containing products
* Abuse of alcohol
* Positive drug test or history of drug abuse

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2017-04-13 (Actual); Study Completion 2017-04-13 (Actual)

PRIMARY OUTCOMES:
assessment of safety data (counts and percentages of adverse events) | Day 0 - Day 28
  counts and percentages of adverse events

SECONDARY OUTCOMES:
Pharmacokinetics (serum concentration of SYNT001) | Pre-dose and 0.08, 2, 4, 6, 8, 12, 16, 20, 24, 48, 72, and 120 hours post dose
  serum concentration of SYNT001
Pharmacodynamics | Days 1 (pre dose), 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 21 and 28
  total serum IgG levels

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No